CLINICAL TRIAL: NCT02057003
Title: Security and Efficacy of Triple Therapy Including Direct-Acting Antivirals Against Chronic Hepatitis C Infection In HIV-Coinfected Patients In Real-Life Conditions: The Prospective HEPAVIR Cohort.
Brief Title: Real-life Security and Efficacy of DAA-based Therapy in HCV/HIV-Coinfected Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Valme University Hospital (Other)
Collaborators: Hospital Universitario Reina Sofia de Cordoba (Other Government); Hospital Universitario Virgen de la Victoria (Other); Fundación de Investigación Biomédica - Hospital Universitario de La Princesa (Other); Hospital Regional de Malaga (Other); Hospital Torrecárdenas (Unknown); Complejo Hospitalario Universitario de Huelva (Other); Hospital Universitario Puerta del Mar (Other); Hospital Universitario Virgen Macarena (Other); Hospital La Línea (Unknown); Complejo Hospitalario de Jaén (Unknown); Hospital Universitario Puerto Real (Other); Hospital Universitario de Canarias (Other); Hospital Poniente (Unknown); Hospital Universitario Central de Asturias (Other); Hospital Álvaro Cunqueiro (Other); Hospital Universitario Virgen de la Arrixaca (Other); Hospital Universitario de Gran Canaria (Unknown)
Responsible Party: Principal Investigator, José A. Mira Escarti, MD, Valme University Hospital
Other Study IDs: HEPAVIR-DAA
Record Dates: First submitted 2014-01-06; First posted 2014-02-06 (Estimated); Last update posted 2016-10-17 (Estimated); Status verified 2016-10

CONDITIONS: Hepatitis C, Chronic; Human Immunodeficiency Virus
Keywords: HIV; hepatitis C virus; sustained virologic response; telaprevir; boceprevir; simeprevir; sofosbuvir; daclatasvir; paritaprevir; pegylated interferon; ribavirin; direct-acting antivirals; dasabuvir; ombitasvir; ledipasvir; velpatasvir; grazoprevir; elbasvir
MeSH Terms: conditions — Hepatitis C, Chronic; Acquired Immunodeficiency Syndrome; Hepatitis C | interventions — telaprevir; N-(3-amino-1-(cyclobutylmethyl)-2,3-dioxopropyl)-3-(2-((((1,1-dimethylethyl)amino)carbonyl)amino)-3,3-dimethyl-1-oxobutyl)-6,6-dimethyl-3-azabicyclo(3.1.0)hexan-2-carboxamide; Simeprevir; Sofosbuvir; daclatasvir; ombitasvir; paritaprevir; dasabuvir; ledipasvir; grazoprevir; elbasvir; velpatasvir

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- DAA-based therapy against HCV: HIV/HCV-coinfected patients who start therapy against HCV including one or more DAA
  Interventions: Drug: DAA against HCV

INTERVENTIONS:
Drug: DAA against HCV
  Other Names: telaprevir; boceprevir; simeprevir; sofosbuvir; daclatasvir; ombitasvir; paritaprevir; dasabuvir; ledipasvir; grazoprevir; elbasvir; velpatasvir

SUMMARY:
The purpose of this study is to evaluate the efficacy and tolerability of DAA-based regimens in the clinical practice in HIV/HCV-coinfected patients.

Hypothesis: The efficacy and tolerability of DAA-based regimens in the clinical practice is different to what is observed in clinical trials in HIV/HCV-coinfected patients.

DETAILED DESCRIPTION:
Treatment strategies aimed to achieve sustained virologic response (SVR) are of highest priority in patients with chronic hepatitis C and HIV coinfection, since SVR leads to a dramatic reduction in the incidence of hepatic decompensations and mortality in this setting. Until recently, therapy against hepatitis C virus (HCV) was based on pegylated interferon (peg-IFN) plus ribavirin (RBV). This combination prompt SVR only in approximately 50% of the HCV genotype 1 (HCV-1)-infected patients. Furthermore, it is costly and associated with multiple and sometimes serious side effects. In the setting of HIV/HCV-1-coinfection, rates of SVR are even lower and do not exceed 25% in the clinical practice.

Considerable increases of SVR have been achieved recently with the arrival of direct acting antivirals (DAA) against HCV. Among the first of these new agents are the protease inhibitors telaprevir (TVR) and boceprevir (BOC), which are approved for HCV-1 infection. Data obtained from clinical trials have demonstrated that the combination of peg-IFN/RBV with TVR or BOC significantly augments SVR rates as compared to what is observed with peg-IFN plus RBV only. As a consequence, triple therapy including peg-IFN, RBV plus TVR or BOC has become the standard therapy for HCV-1-infected patients in our setting. In addition, a number of further DAAs are currently in the final phases of development, as it is the case for the protease inhibitors faldaprevir and simeprevir, the polymerase NS5B inhibitor sofosbuvir and the NS5A inhibitor daclatasvir.

Although the considerable improvement of therapy outcome with DAA-including regimens is giving a positive prospective, there are a number of questions that have to be solved as soon as possible. On the one hand, the information on response to DAA in the coinfected population is derived from clinical trials, which often do not reflect patient management in the clinical practice. Also, the populations included in clinical trials are highly selective and may lack the high proportion of difficult-to-treat individuals expected among the candidate population, i.e., those who failed previous treatment and who bear compensated cirrhosis. In fact, data derived from the French cohort CUPIC including HCV-monoinfected, cirrhotic patients, show that tolerability and efficacy of TVR and BOC-based treatment is lower than observed in pivotal trials. On the other hand, similar to dual therapy including Peg-IFN/RBV, it is possible that both response rates and safety profiles of DAAs are not comparable between HCV-monoinfected and HIV/HCV-coinfected patients. In this context, the coinfected population has singularities as the coadministration of antiretroviral therapy, that may cause drug-drug-interactions and decreased tolerability, thus resulting in diminished efficacy. Finally, it is of highest relevance to identify predictive factors for treatment response in the new DAA-based regimens in order to individualize treatment decision and duration of therapy.

Due to the above mentioned, studies on safety and efficacy of DAA-based therapy under real life conditions in HIV/HCV-coinfected patients are urgently needed.

Primary objectives:

* To determine the efficacy of DAA-based therapy in the clinical in patients with chronic hepatitis C and HIV coinfection.
* To determine the security of DAA-based therapy in the clinical in patients with chronic hepatitis C and HIV coinfection.

Secondary objectives:

* Identification of predictive factors for response to DAA-based treatment in the studied population.
* Compare security and efficacy of the different DAAs used.
* Evaluate the on-treatment HCV kinetics for the different regimens.

Scheduled visits: 0, 1, 2, 4, 8, 12, 24, 36 and 48 weeks, as well as 12 and 24 weeks post-treatment.

Definition SVR: Undetectable HCV-RNA 24 weeks after scheduled end of treatment.

Definition of hepatic fibrosis:

* advanced fibrosis: F3 as determined by liver biopsy or 11 kilopascals as determined by transient elastometry
* cirrhosis: F4 as determined by liver biopsy or 14.6 kilopascals as determined by transient elastometry

Variables collected within in the cohort:

* primary outcome variable: SVR (efficacy study) and % of patients who discontinued therapy due to adverse events (safety study)
* epidemiological variable: age, sex, interleukin 28B rs12979860 genotype
* variables related to hepatitis C virus-infection: infection route, genotype, grade of hepatic fibrosis and method used for its determination, baseline Child-Pough-Index, previous hepatic decompensations
* treatment-related variables: previous response to treatment, doses and dose reductions/discontinuations of peg-IFN, RBV and the DAA(s), overall severe adverse events, adverse events that occur in more than 5% of the patients, hepatic decompensations, deaths, HCV viral load at baseline and at each visit
* variables related to HIV-infection: Centers for Disease Control and Prevention (CDC) category, HIV viral load, cluster of differentiation 4 (CD4) cell count, antiretroviral regimen
* analytical variables: aspartate aminotransferase (AST), alanine aminotransferase (ALT), platelets, leucocytes, low-density lipoprotein cholesterol, bilirubin, gamma-glutamyltransferase (GGT), alkaline phosphatase,
* clinical variables: alcohol intake Quality assurance and data checks: Data will be obtained from controlled databases at the participating centers. Databases will be monitored and controlled by queries every three months. Descriptive statistics will be be applied in order to detect transcription errors.

Source data verification: not planned.

All grade 3 or 4 adverse events, as well as all unexpected events, will be reported to the Andalusian Center for Pharmacovigilance (Centro Andaluz de Farmacovigilancia, www.cafv.es).

A sample size of 230 is planned for this study.

Statistical analysis: The outcome variables of this study will be the achievement of SVR, as well as the development of severe adverse events during follow-up. Descriptive statistical analysis will be performed in order to describe the cohort. Continuous variables will be expressed as median [interquartile range (IQR)] and categorical variables as number [percentage; 95% confidence interval (CI)]. The association of continuous variables with SVR or the frequency of patients who discontinue therapy will be analyzed using the Student's t-test for normal distribution and the Mann-Whitney U-test otherwise whereas the relationship with categorical variables will be determined applying the χ2-test or the Fisher's test, when applicable. Those factors that show an association in the univariate analysis with a p<0.2, as well as those with a biologically possible influence, will be entered logistic regression in order to identify independent predictors for SVR. The adjusted odds ratio (AOR) and the respective 95% CI will be calculated. All p values <0.05 will be considered statistically significant. Data will be analyzed using the SPSS statistical software package release 19.0 (SPSS Inc., Chicago, Illinois, USA) and STATA 9.0 (StataCorp, College Station, Texas, USA).

Sample size calculations: Estimating a SVR rate of 55%, with a confidence interval of 95% and a lost-to-follow-up rate of 5%, a minimum of 230 patients should be included in order to obtain a precision of 5%.

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 years
* HIV infection determined by enzymeimmunoassay and confirmed by Western Blot
* Naïve to treatment including a DAA
* Initiation of triple therapy including a DAA
* Written informed consent to participate in the study and to undergo genetic determinations

Exclusion Criteria:

* Pregnancy
* Any contraindication for the administration of peg-IFN, RBV or the respective DAA
* Patients who are not able to provide informed consent to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who consecutively attend the Unit of Infectious Diseases of the Study Group for Viral Hepatitis (HEPAVIR) of the Andalusian Society of Infectious Diseases (Sociedad Andaluza de Enfermedades Infecciosas, SAEI), Spain, will be considered for this study.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2012-01; Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Number of patients who achieve SVR to DAA-based therapy as measure of efficacy | 18 months
  Achievement of SVR to DAA-based therapy in the clinical practice in patients with chronic hepatitis C and HIV coinfection.
Number of patients who develop severe adverse events as measure of safety | 18 months
  Development of severe adverse events related to DAA-based therapy in the clinical practice in patients with chronic hepatitis C and HIV coinfection.

SECONDARY OUTCOMES:
Number of patients who achieve SVR to a BOC-based regimen as compared to numbers of patients who achieve SVR to a TVR-based regimen. | 18 months
  In order to compare TVR- and BOC-based therapy, the numbers of patients who achieve SVR to DAA-based therapy will be analyzed.
Number of patients who reach undetectable HCV-RNA at week 4 of PI-based therapy as a measure of on-treatment response to therapy. | 18 months
Number of patients who develop adverse events during a BOC-based regimen as compared to numbers of patients who develop adverse events during a TVR-based regimen. | 18 months
  In order to compare TVR- and BOC-based therapy, the numbers of patients who develop adverse events during either treatment will be analyzed.
Number of patients who achieve SVR to an interferon-free regimen. | 36 weeks
  The numbers of patients who achieve SVR to DAA-based therapy in absence of interferon will be analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Karin Neukam, PhD, Principal Investigator — Valme University Hospital
Locations (1):
- Valme University Hospital, Seville, Spain

REFERENCES:
- [Background] Coverdale SA, Khan MH, Byth K, Lin R, Weltman M, George J, Samarasinghe D, Liddle C, Kench JG, Crewe E, Farrell GC. Effects of interferon treatment response on liver complications of chronic hepatitis C: 9-year follow-up study. Am J Gastroenterol. 2004 Apr;99(4):636-44. doi: 10.1111/j.1572-0241.2004.04085.x. PMID 15089895
- [Background] Berenguer J, Alvarez-Pellicer J, Martin PM, Lopez-Aldeguer J, Von-Wichmann MA, Quereda C, Mallolas J, Sanz J, Tural C, Bellon JM, Gonzalez-Garcia J; GESIDA3603/5607 Study Group. Sustained virological response to interferon plus ribavirin reduces liver-related complications and mortality in patients coinfected with human immunodeficiency virus and hepatitis C virus. Hepatology. 2009 Aug;50(2):407-13. doi: 10.1002/hep.23020. PMID 19575364
- [Background] Mira JA, Rivero A, de Los Santos-Gil I, Lopez-Cortes LF, Giron-Gonzalez JA, Marquez M, Merino D, del Mar Viloria M, Tellez F, Rios-Villegas MJ, Omar M, Rivero-Juarez A, Macias J, Pineda JA; Grupo HEPAVIR de la Sociedad Andaluza de Enfermedades Infecciosas (SAEI). Hepatitis C virus genotype 4 responds better to pegylated interferon with ribavirin than genotype 1 in HIV-infected patients. AIDS. 2012 Aug 24;26(13):1721-4. doi: 10.1097/QAD.0b013e3283568884. PMID 22695304
- [Background] Jacobson IM, McHutchison JG, Dusheiko G, Di Bisceglie AM, Reddy KR, Bzowej NH, Marcellin P, Muir AJ, Ferenci P, Flisiak R, George J, Rizzetto M, Shouval D, Sola R, Terg RA, Yoshida EM, Adda N, Bengtsson L, Sankoh AJ, Kieffer TL, George S, Kauffman RS, Zeuzem S; ADVANCE Study Team. Telaprevir for previously untreated chronic hepatitis C virus infection. N Engl J Med. 2011 Jun 23;364(25):2405-16. doi: 10.1056/NEJMoa1012912. PMID 21696307
- [Background] Poordad F, McCone J Jr, Bacon BR, Bruno S, Manns MP, Sulkowski MS, Jacobson IM, Reddy KR, Goodman ZD, Boparai N, DiNubile MJ, Sniukiene V, Brass CA, Albrecht JK, Bronowicki JP; SPRINT-2 Investigators. Boceprevir for untreated chronic HCV genotype 1 infection. N Engl J Med. 2011 Mar 31;364(13):1195-206. doi: 10.1056/NEJMoa1010494. PMID 21449783
- [Background] Hezode C, Fontaine H, Dorival C, Larrey D, Zoulim F, Canva V, de Ledinghen V, Poynard T, Samuel D, Bourliere M, Zarski JP, Raabe JJ, Alric L, Marcellin P, Riachi G, Bernard PH, Loustaud-Ratti V, Metivier S, Tran A, Serfaty L, Abergel A, Causse X, Di Martino V, Guyader D, Lucidarme D, Grando-Lemaire V, Hillon P, Feray C, Dao T, Cacoub P, Rosa I, Attali P, Petrov-Sanchez V, Barthe Y, Pawlotsky JM, Pol S, Carrat F, Bronowicki JP; CUPIC Study Group. Triple therapy in treatment-experienced patients with HCV-cirrhosis in a multicentre cohort of the French Early Access Programme (ANRS CO20-CUPIC) - NCT01514890. J Hepatol. 2013 Sep;59(3):434-41. doi: 10.1016/j.jhep.2013.04.035. Epub 2013 May 10. PMID 23669289
- [Derived] Gonzalez-Serna A, Corma-Gomez A, Tellez F, Corona-Mata D, Rios-Villegas MJ, Merino D, Galera C, Collado-Romacho AR, De Los Santos I, Cucurull J, Santos M, Garcia-Martin S, Rivero A, Real LM, Macias J. Response to glecaprevir/pibrentasvir in HIV/HCV-coinfected patients in clinical practice. J Antimicrob Chemother. 2023 Oct 3;78(10):2591-2596. doi: 10.1093/jac/dkad278. PMID 37671831
- [Derived] Macias J, Morano LE, Tellez F, Granados R, Rivero-Juarez A, Palacios R, Rios M, Merino D, Perez-Perez M, Collado A, Figueruela B, Morano A, Freyre-Carrillo C, Martin JM, Rivero A, Garcia F, Pineda JA; HEPAVIR group from the Sociedad Andaluza de Enfermedades Infecciosas (SAEI) and the GEHEP group from the Sociedad Espanola de Enfermedades Infecciosas y Microbiologia (SEIMC). Response to direct-acting antiviral therapy among ongoing drug users and people receiving opioid substitution therapy. J Hepatol. 2019 Jul;71(1):45-51. doi: 10.1016/j.jhep.2019.02.018. Epub 2019 Mar 8. PMID 30853642